CLINICAL TRIAL: NCT00819182
Title: Breathe-intervention for Hot Flashes, Associated Outcomes, and Interference
Brief Title: Breathe for Hot Flashes Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0803-13; R01CA132927 (NIH)
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Hot Flashes
Keywords: Menopause; Breast Cancer; Hot Flash; Night Sweats
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Paced respiration (Experimental): The paced respiration intervention group received a compact disc with paper booklet. The booklet reinforced instructions on the first audio track for how to accomplish a target breath rate of 6-8 breaths per minute, practice twice per day for 15 minutes, and apply the breathing at the onset of each hot flash. Women were instructed to do slow, deep, abdominal breathing in through the nose and out through the mouth as per international recommendations (4). They were also instructed to practice twice per day for 15 minutes as per the small, laboratory-based studies (5, 6). The second and third tracks contained specially composed, digitally recorded music to help entrain the breath rate and structure the length of practice.
  Interventions: Behavioral: Paced respiration
- Sham comparator: Fast, shallow breathing (Sham Comparator): The sham comparator group received a digital videodisc with paper booklet. The booklet reinforced voice-over and video demonstration to practice twice per day and apply the fast shallow breathing at the onset of each flash. A previously published report provides additional details and data indicating this program was a suitable attention control.
  Interventions: Behavioral: Sham comparator: fast shallow breathing
- Control: Usual Care (No Intervention): The usual care group received an investigator-signed letter explaining they were not selected to receive any study materials during the 16-week follow-up. These participants received paced respiration materials by mail after study completion.

INTERVENTIONS:
Behavioral: Paced respiration — Breathing exercise
  Arms: Paced respiration
Behavioral: Sham comparator: fast shallow breathing — sham breathing exercise
  Arms: Sham comparator: Fast, shallow breathing

SUMMARY:
Background: Paced respiration has been internationally recommended for vasomotor symptom management despite limited empirical evidence.

Objective: To evaluate efficacy of a paced respiration intervention against a sham comparator breathing control and usual care control for vasomotor and other menopausal symptoms.

Design: A 16-week, 3-group, partially blinded, controlled trial with 2:2:1 randomization and stratification by group (breast cancer, no cancer), Midwestern city and surrounding area.

Participants: 218 randomized women (96 breast cancer survivors, 122 menopausal women without cancer) recruited through community mailings and registries.

Interventions: Training, home practice support, and instructions to use the breathing at the time of each hot flash were delivered via compact disc with printed booklet (paced respiration intervention) or digital videodisc with printed booklet (fast shallow breathing control). Usual care control received a letter regarding group assignment.

Main Measures: Hot flash frequency, severity, and bother (primary), hot flash interference in daily life, perceived control over hot flashes, and mood and sleep disturbances (secondary). Intervention performance, adherence, and adverse events were assessed.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Reporting daily hot flashes and desirous of hot flash treatment
* Peri- or post menopausal
* Living within a 60-mile radius of Indianapolis or willing to drive to the center for all study visits
* Able to read, write, and speak English
* in good general health

In addition:

* Breast Cancer survivors will have a known diagnosis of non-metastatic disease
* No history of other cancers
* Be at least four weeks post-completion of surgery, radiation and chemotherapy

Exclusion Criteria:

* Known psychiatric disorders or cognitive impairments
* Participation in our previous pilot study evaluating our control condition
* Self-reported difficulties with normal everyday breathing
* Meet criteria at baseline for number of subjective and/or objective hot flashes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet S Carpenter, PhD, RN, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Nursing, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data available upon request.

REFERENCES:
- [Result] Carpenter JS, Burns DS, Wu J, Otte JL, Schneider B, Ryker K, Tallman E, Yu M. Paced respiration for vasomotor and other menopausal symptoms: a randomized, controlled trial. J Gen Intern Med. 2013 Feb;28(2):193-200. doi: 10.1007/s11606-012-2202-6. PMID 22936289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from April 1, 2009 to February 1, 2011. Participants were recruited by mass mailings to community-dwelling women and registry participants. Additionally, recruitment occurred in breast cancer and high-risk clinics in the Midwest.
Groups:
- Paced Respiration: The paced respiration intervention group received a compact disc with paper booklet. The booklet reinforced instructions on the first audio track for how to accomplish a target breath rate of 6-8 breaths per minute, practice twice per day for 15 minutes, and apply the breathing at the onset of each hot flash. Women were instructed to do slow, deep, abdominal breathing in through the nose and out through the mouth as per international recommendations. They were also instructed to practice twice per day for 15 minutes as per the small, laboratory-based studies. The second and third tracks contained specially composed, digitally recorded music to help entrain the breath rate and structure the length of practice.
- Fast, Shallow Breathing: The fast, shallow comparator group received a digital videodisc with paper booklet. The booklet reinforced voice-over and video demonstration to practice twice per day and apply the fast shallow breathing at the onset of each flash.
- Usual Care: The usual care group received an investigator-signed letter explaining they were not selected to receive any study materials during the 16-week follow-up. These participants received paced respiration materials by mail after study completion.
Period: Overall Study
Arm/Group | Paced Respiration | Fast, Shallow Breathing | Usual Care
Started | 88 (Consented participants allocated to this arm.) | 86 (Consented participants allocated to this arm.) | 44 (Consented participants allocated to this arm.)
Week 16 Visit | 75 | 78 | 43
Completed | 75 | 78 | 43
Not Completed | 13 | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paced Respiration | Fast, Shallow Breathing | Usual Care | Total
Number analyzed (Participants) | 88 | 86 | 44 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.44 (6.84) | 51.93 (6.81) | 53.52 (5.68) | 52.86 (6.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 86 | 44 | 218
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 85 | 86 | 44 | 215
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 23 | 21 | 12 | 56
  White | 61 | 62 | 32 | 155
  More than one race | 2 | 3 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 88 | 86 | 44 | 218
Breast Cancer History [Number; unit: Participants] — Breast cancer survivors > 4 weeks post-completion of surgery, radiation, and/or chemotherapy for nonmetastatic breast cancer with no additional cancer history OR menopausal women with no cancer history
  Participants
    Breast Cancer Survivor | 38 | 38 | 20 | 96
    Menopausal Women with No Cancer History | 50 | 48 | 24 | 122
Hot Flash Frequency [Mean (Standard Deviation); unit: Hot flashes per 24 hr] — Prospective, real-time electronic diary used by participants for a minimum of 24 hours to a maximum of 7 days. Duration of use was determined by participant choice.
  Hot flashes per 24 hr | 7.02 (4.32) | 6.43 (3.96) | 7.31 (4.04) | 6.84 (4.12)
Hot Flash Severity [Mean (Standard Deviation); unit: Scores on a scale] — Self-reported rating using a scale from 0 (not at all severe) to 10 (extremely severe). Calculated as 24 hour averages.
  Scores on a scale | 4.50 (1.60) | 5.23 (1.58) | 5.40 (1.26) | 5.17 (1.53)
Hot Flash Bother [Mean (Standard Deviation); unit: Scores on a scale] — Self-reported rating using a scale from 0 (not at all bothersome) to 10 (extremely bothersome). Calculated as 24 hour averages.
  Scores on a scale | 4.52 (1.72) | 4.78 (1.72) | 4.69 (1.32) | 4.66 (1.64)
Hot Flash Related Daily Interference [Mean (Standard Deviation); unit: Scores on a scale] — Self-report using well-validated, standardized questionnaire. Subject rated interference items on scale from 0 to 10. Total score range was 0-100 with higher scores indicating greater interference with daily life.
  Scores on a scale | 3.99 (2.35) | 4.58 (2.46) | 4.51 (2.61) | 4.32 (2.43)
Perceived Control Over Hot Flashes [Mean (Standard Deviation); unit: Scores on a scale] — Self-report using well-validated, standardized questionnaire composed of 15 items with response option ratings of 1-4. Scores were summed with potential range of 15-60. Lower scores indicated less control over hot flashes; higher scores indicate higher perceived control over hot flashes.
  Scores on a scale | 37.38 (4.68) | 37.48 (5.10) | 37.95 (4.64) | 37.57 (4.80)
Mood Disturbance [Mean (Standard Deviation); unit: Scores on a scale] — Self-report using the well-validated Profile of Mood States-Short Form questionnaire. Six subscales are computed. Total scores are computed using the formula Depression-Dejection + Tension-Anxiety + Anger-Hostility + Fatigue-Inertia + Confusion-Bewilderment + (24 - Vigor-Activity). Total scores range from 0 to 124 with higher scores indicating higher mood disturbance.
  Scores on a scale | 40.08 (24.77) | 47.17 (23.03) | 39.50 (24.47) | 43.03 (23.86)
Sleep Disturbance [Mean (Standard Deviation); unit: Global sleep quality score] — Self-report using the Pittsburgh Sleep Quality Index which is composed of 19-items to assess sleep quality and disturbances during the past week. Scores range from 0-21 with higher scores indicating poorer sleep quality and more sleep disturbance.
  Global sleep quality score | 7.38 (3.23) | 8.59 (3.59) | 8.14 (3.66) | 7.99 (3.50)

OUTCOME MEASURES:

1. Primary Outcome: Hot Flash Frequency
Description: Prospective, real-time electronic diary used by participants for a minimum of 24 hours to a maximum of 7 days. Duration of use was determined by participant choice.
Time Frame: 16 weeks
Population: Analysis based on all randomized participants.
Measure: Mean (Standard Deviation); unit: Hot flashes per 24 hr
Arm/Group | Paced Respiration | Fast, Shallow Breathing | Usual Care
Number analyzed (Participants) | 88 | 86 | 44
Hot flashes per 24 hr | 3.48 (3.45) | 3.95 (4.19) | 4.76 (3.54)

2. Secondary Outcome: Hot Flash Related Daily Interference
Description: Self-report using well-validated, standardized questionnaire. Subject rated interference on scale items from 0 to 10. Total score range was 0-100 with higher scores indicating greater interference with daily life.
Time Frame: 16 weeks
Population: Analysis based on all randomized participants.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Paced Respiration | Fast, Shallow Breathing | Usual Care
Number analyzed (Participants) | 88 | 86 | 44
Scores on a scale | 2.75 (2.19) | 3.41 (2.54) | 3.93 (2.15)

3. Secondary Outcome: Perceived Control Over Hot Flashes
Description: Self-report using well-validated, standardized questionnaire composed of 15 items with response option ratings of 1-4. Scores were summed with potential range of 15-60. Lower scores indicated less control over hot flashes; higher scores indicate higher perceived control over hot flashes.
Time Frame: 16 weeks
Population: Analysis based on all randomized participants.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Paced Respiration | Fast, Shallow Breathing | Usual Care
Number analyzed (Participants) | 88 | 86 | 44
Scores on a scale | 42.67 (4.51) | 42.69 (5.69) | 39.60 (4.73)

4. Secondary Outcome: Mood Disturbance
Description: Self-report using the well-validated Profile of Mood States-Short Form questionnaire. Six subscales are computed. Total scores are computed using the formula Depression-Dejection + Tension-Anxiety + Anger-Hostility + Fatigue-Inertia + Confusion-Bewilderment + (24 - Vigor-Activity). Total scores range from 0 to 124 with higher scores indicating higher mood disturbance.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Paced Respiration | Fast, Shallow Breathing | Usual Care
Number analyzed (Participants) | 88 | 86 | 44
Scores on a scale | 38.26 (25.79) | 40.13 (20.32) | 43.48 (30.37)

5. Secondary Outcome: Sleep Disturbance
Description: Self-report using the Pittsburgh Sleep Quality Index which is composed of 19-items to assess sleep quality and disturbances during the past week. Scores range from 0-21 with higher scores indicating poorer sleep quality and more sleep disturbance.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Global Sleep Disturbance Score
Arm/Group | Paced Respiration | Fast, Shallow Breathing | Usual Care
Number analyzed (Participants) | 88 | 86 | 44
Global Sleep Disturbance Score | 6.81 (3.37) | 7.66 (3.15) | 8.23 (3.82)

6. Primary Outcome: Hot Flash Severity
Description: Self-reported rating using a scale from 0 (not at all severe) to 10 (extremely severe). Calculated as 24 hour averages at 16 week timepoint.
Time Frame: 16 weeks
Population: Analysis based on all randomized participants.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Paced Respiration | Fast, Shallow Breathing | Usual Care
Number analyzed (Participants) | 88 | 86 | 44
Scores on a scale | 4.33 (2.06) | 4.65 (2.07) | 5.20 (1.89)

7. Primary Outcome: Hot Flash Bother
Description: Self-reported rating using a scale from 0 (not at all bothersome) to 10 (extremely bothersome). Calculated as 24 hour averages at 16 week timepoint.
Time Frame: 16 weeks
Population: Analysis based on all randomized participants.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Paced Respiration | Fast, Shallow Breathing | Usual Care
Number analyzed (Participants) | 88 | 86 | 44
Scores on a scale | 3.89 (1.93) | 4.22 (2.19) | 4.76 (1.73)

8. Other Pre Specified Outcome: Intervention Performance
Description: Physiological recordings of number of breaths per minute to verify correct performance of paced respiration for this participant group only. Assessment was conducted in a single visit scheduled 2 weeks post-randomization for the paced respiration group.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Breaths Per Minute
Arm/Group | Paced Respiration
Number analyzed (Participants) | 88
Breaths Per Minute | 7.35 (2.45)

9. Other Pre Specified Outcome: Intervention Performance
Description: Physiological recordings of number of breaths per minute to verify correct performance of paced respiration for this participant group only. Assessment was conducted at the week 16 post-randomization timepoint.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Breaths Per Minute
Arm/Group | Paced Respiration
Number analyzed (Participants) | 88
Breaths Per Minute | 6.97 (1.92)

10. Other Pre Specified Outcome: Intervention Adherence
Description: Number of breathing practice sessions per participant over the 16 week study period.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Total practice sessions in 16 weeks
Arm/Group | Paced Respiration | Fast, Shallow Breathing
Number analyzed (Participants) | 88 | 86
Total practice sessions in 16 weeks | 109.83 (67.76) | 133.93 (78.27)

ADVERSE EVENTS:
Arm/Group | Paced Respiration | Fast, Shallow Breathing | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/86 | 0/44
Other Adverse Events (participants affected / at risk) | 0/88 | 0/86 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No